CLINICAL TRIAL: NCT06253247
Title: Effect of NanoChitosan Impregnated Calcium Hydroxide Paste as an Intracanal Medication on the Intensity of Postoperative Pain and Bacterial Load Reduction in Necrotic Teeth: A Randomized Controlled Trial
Brief Title: Effect of NanoChitosan Impregnated Calcium Hydroxide as an Intracanal Medication on Postoperative Pain Intensity and Bacterial Load Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Osama ElGhannam, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICM 101
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Intervention

STUDY DESIGN:
Intervention Model Description: Parallel randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors (patients and statistician) will not know which group the participants are related to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with necrotic mandibular premolars will be treated with NanoChitosan impregnated Ca(OH)2 (Experimental): 25-45 years old patients with necrotic single rooted mandibular premolars with single canal will be treated with NanoChitosan impregnated Calcium Hydroxide as an intracanal medicament for 7 days
  Interventions: Combination Product: NanoChitosan impregnated Calcium Hydroxide
- Patients with necrotic mandibular premolars will be treated with Calcium Hydroxide (Active Comparator): 25-45 years old patients with necrotic single rooted mandibular premolars with single canal will be treated with calcium hydroxide as an intracanal medicament for 7 days
  Interventions: Combination Product: NanoChitosan impregnated Calcium Hydroxide

INTERVENTIONS:
Combination Product: NanoChitosan impregnated Calcium Hydroxide — NanoChitosan impregnated Calcium Hydroxide used as an intracanal medication fro 7 days

SUMMARY:
This research will study the effect of NanoChitosan impregnated Calcium Hydroxide versus Calcium Hydroxide as an intracanal medication on postoperative pain intensity measured using numerical rating scale (NRS) and bacterial load reduction determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml) in necrotic teeth.

DETAILED DESCRIPTION:
Primary outcome: Postoperative pain measured using numerical rating scale (NRS)

1. After placement of intracanal medicament at 6, 12, 24 and 48 hours.
2. After root canal obturation at 6, 12, 24 and 48 hours.

Secondary outcome: Bacterial load reduction determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml)

1. Sample 1 (S1): after access preparation and pre-instrumentation.
2. Sample 2 (S2): post-instrumentation.
3. Sample 3 (S3): post-intracanal medicament removal at 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25-45 years old.
2. Males or females.
3. Healthy patients who are categorized as I or II according to The American Society of Anesthesiologists. (ASA I or II)
4. Patients' accepting to participate in the trial.
5. Patients who can understand the pain scale and can sign the informed consent.
6. Mandibular Single rooted premolars, having single root canal: Diagnosed clinically with pulp necrosis.
7. Positive pain on percussion denoting apical periodontitis.(20)
8. Slight widening in the periodontal membrane space
9. Normal occlusal contact with opposing teeth

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders (ASA III or IV).
2. If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively.
3. Pregnant women
4. Patients reporting bruxism, clenching, TMJ problems or traumatic occlusion
5. Patients with two or more adjacent teeth requiring endodontic treatment.
6. Teeth that require further procedural steps or multidisciplinary approach.

   1. Association with swelling or fistulous tract.
   2. Acute periapical abscess.
   3. Mobility Grade II or III.
   4. Pocket depth more than 5mm.
   5. Previous root canal treatment.
   6. Non-restorable.
   7. Immature root.
   8. Radiographic evidence of external or internal root resorption, vertical root fracture, perforation, calcification.
7. Inability to perceive the given instructions.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measured using numerical rating scale | 48 hours
  postoperative pain will be recorded after placement of intracanal medicament and after root canal obturation using numerical rating scale ,An 11-point scale from 0-10 representing pain intensity ,"10" being the most intense pain conceivable.

SECONDARY OUTCOMES:
Bacterial load reduction | T0=Baseline immediate after access preparation . T1=Post-instrumentation. T2=post-intracanal medicament removal at 7 days.
  Bacterial load reduction determined by bacterial counting using agar culture technique after root canal preparation (Number of colony forming unit per millilitre)
Incidence of inter- appointment flare up | Up to 48 hours post- operatively
  recording the incidence of inter-appointment flare up with a binary scale
Number of analgesic tablets taken by the patient after endodontic treatment | Up to 48 hours post- operatively
  Number of analgesic tablets intake after root canal treatment, using numerical counting.

IPD SHARING:
Plan to Share IPD: Yes